CLINICAL TRIAL: NCT03674554
Title: Prosthetic Complications of Screw Retained Restoration Using Multi-unit Abutments Versus Intra-oral Luting on Titanium Base in Implant Supported Complete Overdentures Randomized Clinical Trial
Brief Title: Prosthetic Complications of Screw Retained Restoration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mostafa said hosny, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 28809010109913
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Edentulous Jaw; Edentulous Alveolar Ridge; Edentulous Mouth
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation sequence generation will be performed by the Senior supervisor. Enrolment of participants will be performed by the principle investigator where the patients will be assessed for eligibility.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- titanium bases group (Experimental): full-arch screw-retained implant prosthesis on titanium bases using intra oral luting cement technique
  Interventions: Procedure: titanium bases using intra oral luting cement technique
- transmucosal abutment group (Experimental): a full-arch screw-retained implant prosthesis with transmucosal abutment
  Interventions: Procedure: transmucosal abutment

INTERVENTIONS:
Procedure: titanium bases using intra oral luting cement technique — a full-arch screw-retained implant prosthesis on titanium bases using intra oral luting cement technique
  Arms: titanium bases group
Procedure: transmucosal abutment — a full-arch screw-retained implant prosthesis with transmucosal abutment
  Arms: transmucosal abutment group

SUMMARY:
On of the main fixed prosthetic options of completely edentulous patients is the screw-retained implant supported prosthesis which was constructed on transmucosal abutments with its encountered problems such as: hardness to make it passively seated with multiple screw fracture and loosening problems and multiple encountered veneer material fracture and so there effect on patient satisfaction with multiple maintenance recalls.so, the investigators want to try a new technique of fabrication which was proposed for reducing the problems of lack of passivity which is the intraoral luting cement technique on titanium bases with reduced screw number but, with luting cement problems as de-cementation and cement biological effects on soft tissues and bone and there effect on number of patient recall visits and maintenance and so there effect on patient satisfaction

ELIGIBILITY:
Inclusion Criteria:

* - Completely edentulous patients
* Patients with completely edentulous ridges have an opposing natural dentition or implant supported overdenture
* Completely edentulous patients (with the above mentioned criteria) who have proper amount of attached gingiva (≥2 mm) or to be created
* Completely edentulous patients (with the above mentioned criteria) who have no history of bruxism
* Completely edentulous patients (with the above mentioned criteria) who were free or controlled diabetic assessed by measuring glycosylated haemoglobin (HbA1c). (lesser than or equal to 6.4 percent )

Exclusion Criteria:

* - Patients having a medical condition that absolutely contraindicates implant placement.
* Patients with uncontrolled diabetes, assessed by measuring glycosylated haemoglobin (HbA1c). (greater than to 6.4 percent )
* Potentially uncooperative patients who are not willing to go through the proposed interventions. - Moderate-to-heavy daily smokers* (who report consuming at least 11 cigarettes/day).
* Patients who are having complete lower denture
* Patients who have history of bruxism

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Abutment screw loosening | 12 months
  Measuring device :Clinical visual inspection / Measuring unit:Binary

SECONDARY OUTCOMES:
Prosthetic screw loosening | 12 months
  Measuring device :Clinical visual inspection / Measuring unit:Binary
Prosthetic screw fracture | 12 months
  Measuring device :Clinical visual inspection / Measuring unit:Binary
Abutment screw fracture | 12 months
  Measuring device :Clinical visual inspection / Measuring unit:Binary
Veneer fracture | 12 months
  Measuring device :Clinical visual inspection / Measuring unit:Binary
Framework fracture | 12 months
  Measuring device :Clinical visual inspection / Measuring unit:Binary
Ti-bases de-cementation | 12 months
  Measuring device :Clinical visual inspection / Measuring unit:Binary

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Universty, Cairo, Egypt